CLINICAL TRIAL: NCT02940145
Title: Modifications to Phase Angle After Resistance Training Are Associated With Changes in Body Composition, Inflammatory and Oxidative Stress Biomarkers in Older Women
Brief Title: Phase Angle and Body Composition, Inflammatory and Oxidative Stress Biomarkers.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Estadual de Londrina (Other)
Responsible Party: Principal Investigator, Crisieli Maria Tomeleri, Doctor, Universidade Estadual de Londrina
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: UEL09167-1/2014
Record Dates: First submitted 2016-10-17; First posted 2016-10-20 (Estimated); Last update posted 2017-06-20 (Actual); Status verified 2017-06

CONDITIONS: Body Composition, Beneficial; Oxidative Stress; Acute and Chronic Inflammation
Keywords: inflammatory biomarkers; Interleukines; resistance training; phase angle; oxidative stress
MeSH Terms: conditions — Glucocorticoid Receptor Deficiency | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- intervention 1 (Experimental): The training group performed the resistance training (RT) program. All participants were personally supervised by physical education professionals with substantial RT experience. The sessions were performed 3 times per week on Mondays, Wednesdays, and Fridays, wirh 3 sets of 10-15 repetition maximums.The RT program was performed in the following order: chest press, seated row, triceps pushdown, preacher curl, horizontal leg press, knee extension, leg curl, , and seated calf raise.
  Participants were afforded a 1 to 2 min rest interval between sets and 2 to 3 min between each exercise. The training load was consistent with the prescribed number of repetitions for the three sets of each exercise
  Interventions: Other: Resistance Training
- control group (No Intervention): The control group did not perform any type of physical exercise during the intervention period.

INTERVENTIONS:
Other: Resistance Training — The investigation was carried out over a period of 16 weeks, with 12 weeks dedicated to the RT program and 4 weeks allocated for measurements. Anthropometric, body composition, and blood samples measurements were performed at weeks 1-2, and 15-16. A supervised progressive RT was performed between weeks 3-14. The CG did not perform any type of physical exercise during this period.
  Arms: intervention 1

SUMMARY:
The main purpose of the present study was to investigate the effects of 12 weeks of resistance training (RT) on phase angle (PhA), body composition, inflammatory and oxidative stress biomarkers, in older women and to evaluate whether RT induced adaptations on body composition, inflammatory and oxidative stress biomarkers are related to healthy adaptations in PhA.

DETAILED DESCRIPTION:
The investigation was carried out over a period of 16 weeks, with 12 weeks dedicated to the RT program and 4 weeks allocated for measurements. Anthropometric, body composition, and blood samples measurements were performed at weeks 1-2, and 15-16. A supervised progressive RT was performed between weeks 3-14. The CG did not perform any type of physical exercise during this period.

Recruitment was carried out through newspaper and radio advertisings, and home delivery of leaflets in the central area and residential neighborhoods. All participants completed health history and physical activity questionnaires and met the following inclusion criteria: 60 years old or more, physically independent, free from cardiac or orthopedic dysfunction, not receiving hormonal replacement therapy, and not performing any regular physical exercise more than once a week over the six months preceding the beginning of the investigation. After individual interviews, 59 volunteers were dismissed as potential candidates because they did not meet the inclusion criteria for the investigation. The remaining 51 older women were randomly divided into one of two groups: a training group that performed the RT program or a control group that did not perform any type of physical exercise. Anthropometric, body composition (DXA), phase angle, total body water (intra and extracellular water compartments; Xitron 4200 Bioimpedance Spectrum Analyzer), muscular strength (1RM), and blood sample measurements were performed pre- and post-training. Two-way analysis of variance for repeated measures was applied for intra- and inter-group comparisons. When an F-ratio was significant, Fisher's post hoc test was employed to identify mean differences. The statistical power was determined to verify the statistical power of the analysis. Pearson's correlation was used to evaluate the correlation between delta percent changes in body composition, and muscular strength, inflammatory and oxidative stress biomarkers (independent variables) with the percentage change in PhA (dependent variables). Subsequently, linear regression (bivariate analyses) was performed for all variables that presented P<0.05 in the Pearson's correlation analyses. For the multiple comparison the multivariate regression model was performed. For all statistical analyses, significance was accepted at P<0.05.

ELIGIBILITY:
Inclusion Criteria:

* 60 years old or more, physically independent, free from cardiac or orthopedic dysfunction, not receiving hormonal replacement therapy, and not performing any regular physical exercise more than once a week in the six months preceding the beginning of the investigation.
* Participants passed a diagnostic graded exercise stress test with a 12-lead electrocardiogram, reviewed by a cardiologist, and were released with no restrictions for participation in this investigation.

Exclusion Criteria:

• All subjects not participating in 85% of the total sessions of training or withdrawl

Min Age: 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2014-03; Primary Completion 2015-03 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Change in Phase Angle | baseline and 12 weeks
  Spectral bioelectrical impedance device (Xitron Hydra, model 4200, Xitron Technologies, San Diego, CA, USA) was used to estimate the resistance (R), and reactance (Xc), and subsequently the PhA was calculated as arc-tangent (Xc/R) x 180°/π. The results are presented in degree
Change in body composition | baseline and 12 weeks
  Whole-body dual-energy X-ray absorptiometry (DXA) (Lunar Prodigy, model NRL 41990, GE Lunar, Madison, WI) was used to assess body fat, trunk fat and appendicular lean soft tissue. The total skeletal muscle mass (SMM) was estimated by the predictive equation proposed by Kim et al. (Kim et al., 2002). The results are presented in kg.
Change in CRP | baseline and 12 weeks
  Measurements of serum levels of high-sensitivity CRP were carried out using a biochemical auto-analyzer system (Dimension RxL Max - Siemens Dade Behring) according to established methods in the literature consistent with the manufacturer's recommendations. The results are presented in milligrams per decilitre (mg/dL).
Change in cellular hydration | baseline and 12 weeks
  Spectral bioelectrical impedance device (Xitron Hydra, model 4200, Xitron Technologies, San Diego, CA, USA) was used to estimate the intracellular water (ICW), extracellular water (ECW), and total body water (TBW). The results are presented in liters (L)
Change in inflammatory markers | Baseline and 12 weeks
  TNF-α, and IL-6, IL-10 were determined by enzyme-linked immunosorbent assay (ELISA), according to the speciﬁcations of the manufacturer (Quantikine High Sensitivity Kit, R&D Systems, Minneapolis, MN) and performed in a microplate reader Perkin Elmer, model EnSpire (Waltham, MA, USA). All samples were determined in duplicate to guarantee the precision of the results. The results are presented in picograms per milliliter (pg/ml).
Change in CATALASE (CAT) | Baseline and 12 weeks
  The CAT analysis is by measuring the decay in concentration of H2O2, and oxygen generation using the technique described by literature. The reading of the CAT reaction was carried out in a spectrophotometer, ThermoSpectronic® brand, model HELIOS-α (Waltham, MA, USA) at a wavelength of 240 nm. Results are expressed in U / mgHb .
Change in superoxide dismutase (SOD) | Baseline and 12 weeks
  The SOD activity in erythrocytes was determined using the pyrogallol method described by literature. The reading of SOD reaction is performed in a spectrophotometer, ThermoSpectronic® brand, model HELIOS-α (Waltham, MA, USA) at a wavelength of 420 nm. Results are expressed in U / mgHb (Marklund S)
Change in advanced oxidation protein products (AOPP) | Baseline and 12 weeks
  For measurements, advanced oxidation protein products (AOPP) were determined in the plasma using a semiautomatic method. AOPP concentrations were expressed as micromoles per liter (μmol/L) of chloramines-T equivalents.

SECONDARY OUTCOMES:
change in Muscular strength | baseline and 12 weeks
  Maximal dynamic strength was evaluated using the 1RM test assessed on chest press, knee extension, and preacher curl exercises performed in this exact order. Testing for each exercise was preceded by a warm-up set (6-10 repetitions), with approximately 50% of the estimated load used in the first attempt of the 1RM. This warm-up was also used to familiarize the subjects with the testing equipment and lifting technique. The testing procedure was initiated 2 minutes after the warm-up. The subjects were instructed to try to accomplish two repetitions with the imposed load in three attempts in both exercises. The rest period was 3 to 5 min between each attempt, and 5 min between exercises. The 1RM was recorded as the last resistance lifted in which the subject was able to complete only one single maximal execution
Dietary intake | baseline and 12 weeks
  Participants were instructed by a dietitian to complete a food record on three nonconsecutive days (two week days and one weekend day) pre- and post-intervention. Participants were given specific instructions regarding the recording of portion sizes and quantities to identify all food and fluid intake, in addition to viewing food models in order to enhance precision. Total energy intake, protein, carbohydrate, and lipid content were calculated using nutrition analysis software (Avanutri Processor Nutrition Software, Rio de Janeiro, Brazil; Version 3.1.4). All participants were asked to maintain their normal diet throughout the investigation period.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Garber CE, Blissmer B, Deschenes MR, Franklin BA, Lamonte MJ, Lee IM, Nieman DC, Swain DP; American College of Sports Medicine. American College of Sports Medicine position stand. Quantity and quality of exercise for developing and maintaining cardiorespiratory, musculoskeletal, and neuromotor fitness in apparently healthy adults: guidance for prescribing exercise. Med Sci Sports Exerc. 2011 Jul;43(7):1334-59. doi: 10.1249/MSS.0b013e318213fefb. PMID 21694556
- [Background] Kim J, Wang Z, Heymsfield SB, Baumgartner RN, Gallagher D. Total-body skeletal muscle mass: estimation by a new dual-energy X-ray absorptiometry method. Am J Clin Nutr. 2002 Aug;76(2):378-83. doi: 10.1093/ajcn/76.2.378. PMID 12145010
- [Background] Stobaus N, Pirlich M, Valentini L, Schulzke JD, Norman K. Determinants of bioelectrical phase angle in disease. Br J Nutr. 2012 Apr;107(8):1217-20. doi: 10.1017/S0007114511004028. Epub 2011 Sep 28. PMID 22309898
- [Background] Sardinha LB, Lohman TG, Teixeira PJ, Guedes DP, Going SB. Comparison of air displacement plethysmography with dual-energy X-ray absorptiometry and 3 field methods for estimating body composition in middle-aged men. Am J Clin Nutr. 1998 Oct;68(4):786-93. doi: 10.1093/ajcn/68.4.786. PMID 9771855